CLINICAL TRIAL: NCT00581555
Title: A Randomized Pilot Study Evaluating the Efficacy and Safety of Etanercept in Patients With Moderate to Severe Plaque Psoriasis After Cessation of Ciclosporin Therapy
Brief Title: Evaluation of Etanercept in Patients With Plaque Psoriasis After Stopping Ciclosporin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A6-410
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- etanercept (Experimental): Participants were administered a 50 mg dose of etanercept subcutaneously once a week after an initial course of ciclosporin.
  Interventions: Drug: Etanercept
- placebo (Placebo Comparator): Participants were administered placebo subcutaneously once a week after an initial course of ciclosporin.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg QW initiated during taper of ciclosporin
  Other Names: Enbrel
  Arms: etanercept
Other: Placebo — Randomized to placebo during taper of ciclosporin
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the use of etanercept as a replacement therapy for ciclosporin in patients with plaque psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of etanercept as a replacement therapy for ciclosporin in patients with moderate to severe plaque psoriasis who have achieved an adequate response with ciclosporin.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18 and 70 years
* Active and stable plaque psoriasis with a BSA≥10 or PASI≥10.

Exclusion Criteria:

* Evidence of skin conditions other than psoriasis
* Psoralen plus psoralen + ultraviolet A (PUVA), ciclosporin, acitretin, alefacept, anakinra, or any other systemic anti-psoriasis therapy or disease-modifying antirheumatic drugs (DMARD) with 28 days of screening
* ultraviolet B (UVB) therapy, topical steroids, topical Vitamin A or D analog preparations, or anthralin
* Prior exposure to any TNF-inhibitor. Prior exposure to efalizumab
* Corticosteroid dose of prednisone >10 mg/day
* Serious infection
* Receipt of any live vaccine
* Abnormal hematology or chemistry
* Body mass index (BMI) > 38
* Pregnancy or Breastfeeding
* Significant concurrent medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Micali G, Wilsmann-Theis D, Mallbris L, Gallo G, Marino V, Brault Y, Germain JM. Etanercept reduces symptoms and severity of psoriasis after cessation of cyclosporine therapy: results of the SCORE study. Acta Derm Venereol. 2015 Jan;95(1):57-61. doi: 10.2340/00015555-1845. PMID 24682319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Etanercept
Started | 62 | 58
Completed | 19 | 38
Not Completed | 43 | 20
Not completed — Adverse Event | 4 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 18 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other reasons | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etanercept | Total
Number analyzed (Participants) | 62 | 58 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 41.50 (12.97) | 41.78 (9.86) | 41.63 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 45 | 38 | 83
PASI score [Mean (Standard Deviation); unit: units on scale] — Psoriasis Area and Severity Index (PASI) score: range: 0 (none) to 72 (maximum). Body was divided into head, upper extremities, trunk and lower extremities; each area score was combined for final PASI. For each section, percent area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: (erythema, induration, and desquamation); scale: 0 (none) to 4 (maximum). Final PASI= sum of severity parameters for each section times area score times weight of section (head: 0.1, upper extremities: 0.2, trunk: 0.3, lower extremities: 0.4).
  units on scale | 19.35 (6.98) | 20.19 (7.76) | 19.74 (7.26)
PGA [Mean (Standard Deviation); unit: units on scale] — Physician Global Assessment (PGA) score is based on dermatologist's assessment of disease averaged over all lesions. Overall lesions were graded for individual scores of induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease.
  units on scale | 4.07 (0.73) | 4.25 (0.85) | 4.15 (0.78)
DLQI score [Mean (Standard Deviation); unit: units on scale] — Dermatology Life Quality Index (DLQI) is the dermatology-specific quality of life measure used for psoriatic population. The 10 item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
  units on scale | 11.26 (6.30) | 11.20 (7.22) | 11.23 (6.72)

OUTCOME MEASURES:

1. Secondary Outcome: PASI Area Under the Curve (AUC) Between Randomization and Week 24
Description: PASI AUC = Area under the curve from randomization (Week 6) to Week 24.
Time Frame: Randomization to Week 24.
Population: ITT population: included all randomized participants. n equals number of participants with evaluable data.
Measure: Mean (Standard Error); unit: scores on a scale * weeks
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 62 | 58
scores on a scale * weeks
  Week 8 (n= 59, 56) | 20.7 (5.2) | 20.7 (5.4)
  Week 10 (n= 55, 55) | 7.0 (5.3) | 5.0 (5.4)
  Week 12 (n= 52, 55) | 6.7 (5.3) | 4.4 (5.4)
  Week 16 (n= 45, 49) | 17.5 (5.4) | 10.8 (5.4)
  Week 20 (n= 29, 45) | 33.6 (5.6) | 17.5 (5.5)
  Week 24 (n= 21,40) | 54.8 (5.8) | 24.3 (5.5)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 8; Test type: Superiority or Other; p = 0.999, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was covariate; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-14.7 to 14.7], Standard Error of Mean 7.5
Statistical Analysis 2: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 10; Test type: Superiority or Other; p = 0.795, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was covariate; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-12.8 to 16.7], Standard Error of Mean 7.5
Statistical Analysis 3: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 12; Test type: Superiority or Other; p = 0.758, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was covariate; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-12.5 to 17.1], Standard Error of Mean 7.6
Statistical Analysis 4: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 16; Test type: Superiority or Other; p = 0.381, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was covariate; Mean Difference (Final Values) = 6.7, 95% CI 2-sided [-8.3 to 21.6], Standard Error of Mean 7.6
Statistical Analysis 5: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 20; Test type: Superiority or Other; p = 0.041, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 16.1, 95% CI 2-sided [0.8 to 31.4], Standard Error of Mean 7.8
Statistical Analysis 6: Comparison: Placebo vs Etanercept; Analysis at randomization to Week 24; Test type: Superiority or Other; p < 0.001, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was covariate; Mean Difference (Final Values) = 30.5, 95% CI 2-sided [14.8 to 46.3], Standard Error of Mean 8.0

2. Secondary Outcome: Change From Randomization in PGA Score to Week 24
Description: PGA score is based on dermatologist's assessment of disease averaged over all lesions. Overall lesions were graded for individual scores of induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Change = PGA at Week 24 - PGA at baseline.
Time Frame: Randomization to Week 24.
Population: ITT population: included all randomized participants. n equals number of participants with evaluable data for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 21 | 40
scores on a scale | 0.9 [0.4 to 1.3] | 0.2 [-0.2 to 0.6]
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from randomization to Week 24; Test type: Superiority or Other; p = 0.049, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.0 to 1.2], Standard Error of Mean 0.3

3. Secondary Outcome: Relapse (Loss of 50% Improvement in PASI) During the 24 Weeks After Randomization
Description: Relapse was defined as the loss of 50% improvement in PASI.
Time Frame: Randomization to Week 24.
Population: ITT population: that included all randomized participants. n equals number of participants with evaluable data for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 62 | 58
Percentage of participants | 63.77 | 36.23
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from randomization to Week 24; Test type: Superiority or Other; p = 0.002, Pearson chi-square — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors with a logit link, a binomial distribution and an auto-regressive correlation structure

4. Secondary Outcome: Probability of Being Relapse Free During the 24 Weeks After Randomization
Description: Relapse was defined as loss of 50% improvement in PASI. The time to relapse was estimated using a Kaplan-Meier analysis.
Time Frame: Randomization to Week 24.
Population: as for outcome 2
Measure: Number; unit: probability of relapse free
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 62 | 58
probability of relapse free
  Week 4 | 0.93 | 0.91
  Week 8 | 0.84 | 0.84
  Week 12 | 0.44 | 0.69
  Week 16 | 0.34 | 0.60
  Week 20 | 0.22 | 0.58
  Week 24 | 0.17 | 0.58
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority or Other; p = 0.0003, Log Rank; Time to first relapse was estimated using the Kaplan-Meier's, and comparisons between groups was performed using log rank tests

5. Primary Outcome: Change From Randomization in PASI Score to Week 24 (Week 18 of Etanercept Monotherapy/Placebo)
Description: PASI score: range: 0 (none) to 72 (maximum). Body was divided into head, upper extremities, trunk and lower extremities; each area score was combined for final PASI. For each section, percent area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: (erythema, induration, and desquamation); scale: 0 (none) to 4 (maximum). Final PASI= sum of severity parameters for each section times area score times weight of section (head: 0.1, upper extremities: 0.2, trunk: 0.3, lower extremities: 0.4). Change = PASI at Week 24 - PASI at baseline.
Time Frame: Randomization to Week 24.
Population: Intent-To-Treat (ITT) population: included all randomized participants. n equals number of participants with evaluable data for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 21 | 40
scores on a scale | 2.9 [1.0 to 4.8] | -1.8 [-3.5 to -0.0]
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from randomization to Week 24; Test type: Superiority or Other; p < 0.001, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [2.1 to 7.3], Standard Error of Mean 1.3

6. Secondary Outcome: Percent (%) Change of PASI Score From Randomization to Week 24
Description: Percent improvement in PASI score was calculated from Week 6 to Week 24.
Time Frame: Randomization to Week 24.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 19 | 38
percent change | 121.9 [59.9 to 183.9] | -13.3 [-68.4 to 41.8]
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from randomization to Week 24; Test type: Superiority or Other; p = 0.001, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 135.2, 95% CI 2-sided [52.3 to 218.1], Standard Error of Mean 42.3

7. Secondary Outcome: Change From Randomization in DLQI to Week 24
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Randomization to Week 24.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 20 | 40
scores on a scale | 2.0 [-0.4 to 4.3] | -0.4 [-2.5 to 1.7]
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from randomization to Week 24; Test type: Superiority or Other; p = 0.139, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 2.4, 95% CI [-0.8 to 5.5], Standard Error of Mean 1.6

8. Secondary Outcome: DLQI at Each Visit From Baseline
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10 item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Baseline to Week 24.
Population: ITT population: included all randomized participants. n equals number of participants with evaluable data
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 62 | 58
scores on a scale
  Week 2 (n= 28, 30) | 4.1 (0.9) | 4.0 (0.9)
  Week 4 (n= 25, 22) | 3.0 (0.9) | 4.0 (0.9)
  Week 6 (n= 8, 3) | 1.5 (1.2) | 1.9 (1.9)
  Week 8 (n= 58, 55) | 1.6 (0.6) | 1.6 (0.7)
  Week 10 (n= 56, 54) | 1.7 (0.6) | 1.0 (0.7)
  Week 12 (n= 52, 54) | 2.0 (0.7) | 1.0 (0.7)
  Week 16 (n= 44, 48) | 5.5 (0.7) | 2.8 (0.7)
  Week 20 (n= 29, 44) | 6.2 (0.8) | 3.3 (0.7)
  Week 24 (n= 20, 40) | 6.1 (10.9) | 3.6 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 2; Test type: Superiority or Other; p = 0.956, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.3 to 2.5], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 4; Test type: Superiority or Other; p = 0.41, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.6 to 1.5], Standard Error of Mean 1.3
Statistical Analysis 3: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 6; Test type: Superiority or Other; p = 0.844, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-4.8 to 3.9], Standard Error of Mean 2.2
Statistical Analysis 4: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 8; Test type: Superiority or Other; p = 0.968, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.8 to 1.8], Standard Error of Mean 0.9
Statistical Analysis 5: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 10; Test type: Superiority or Other; p = 0.441, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.1 to 2.5], Standard Error of Mean 0.9
Statistical Analysis 6: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 12; Test type: Superiority or Other; p = 0.3, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.9 to 2.8], Standard Error of Mean 0.9
Statistical Analysis 7: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 16; Test type: Superiority or Other; p = 0.008, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [0.7 to 4.5], Standard Error of Mean 1.0
Statistical Analysis 8: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 20; Test type: Superiority or Other; p = 0.005, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [0.9 to 5.0], Standard Error of Mean 1.0
Statistical Analysis 9: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 24; Test type: Superiority or Other; p = 0.031, mixed model of ANCOVA — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; Treatment groups and visits were fixed factors, participant was a random factor and baseline was a covariate; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.2 to 4.6], Standard Error of Mean 1.1

9. Secondary Outcome: Percentage of Rebound Effects
Description: Rebound effects was defined as worsening of psoriasis to 125% of the baseline PASI or appearance of psoriasis variants such as erythrodermic or pustular psoriasis within 12 weeks of discontinuation of therapy.
Time Frame: Baseline to Week 24.
Population: ITT population: included all randomized participants.n equals number of participants with evaluable data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 62 | 58
percentage of participants | 26.67 | 0.00
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Analysis from baseline to Week 24; Test type: Superiority or Other; p = 0.1196, Pearson chi-square or Fisher exact test — P-values were not adjusted for multiplicity and the priori threshold for statistical significance was 0.05; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Arm/Group | Placebo | Etanercept
Serious Adverse Events (participants affected / at risk) | 1/62 | 2/58
Other Adverse Events (participants affected / at risk) | 48/62 | 43/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Etanercept (N=58)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Etanercept (N=58)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Oedema peripheral (Cardiac disorders) | 1 | 0
Inborn error of bilirubin metabolism (Congenital, familial and genetic disorders) | 0 | 1
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Diarrhoea infectious (Gastrointestinal disorders) | 0 | 1
Dysentery (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 1
Gingival hyperplasia (Gastrointestinal disorders) | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 13 | 7
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Throat irritation (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 5
Feeling hot (General disorders) | 2 | 1
Feeling of body temperature change (General disorders) | 2 | 0
Hyperpyrexia (General disorders) | 1 | 0
Injection site anaesthesia (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 2
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Ascariasis (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 13 | 11
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 2
Superinfection (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood cholesterol abnormal (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 4
Blood magnesium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 3
Transaminases increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 5
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 21 | 17
Hyperaesthesia (Nervous system disorders) | 1 | 0
Insomnia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 10 | 3
Presyncope (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Vertigo (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Somatoform disorder (Psychiatric disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renovascular hypertension (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia effluvium (Skin and subcutaneous tissue disorders) | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Herpes simplex (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Injection site dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Injection site rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Tooth repair (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 2 | 1
Hot flush (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 9 | 9
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Migraine with aura (Vascular disorders) | 1 | 0
Secondary hypertension (Vascular disorders) | 2 | 1
Systolic hypertension (Vascular disorders) | 1 | 0
Venous injury (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.